CLINICAL TRIAL: NCT02476019
Title: A Double Blind, Randomized, Placebo-controlled, Single Center, Phase 2a Study to Determine the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of ISIS 463588 (ISIS-FGFR4RX, an Antisense Inhibitor of Fibroblast Growth Factor Receptor 4) Administered Subcutaneously Once Weekly for 13 Weeks in Obese Patients
Brief Title: A Safety, Tolerability, PK, and PD Study of Once Weekly ISIS-FGFR4RX SC in Obese Patients
Acronym: FGFR4-CS2
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Ionis Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ISIS 463588-CS2; NCT02463240 (obsolete NCT alias)
Record Dates: First submitted 2015-06-15; First posted 2015-06-19 (Estimated); Last update posted 2018-06-25 (Actual); Status verified 2018-06

CONDITIONS: Obesity
Keywords: Obesity; Energy Expenditure
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- ISIS-FGFR4RX (Experimental): ISIS-FGFR4RX administered subcutaneously
  Interventions: Drug: ISIS-FGFR4RX
- Placebo (Placebo Comparator): Placebo administered subcutaneously
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: ISIS-FGFR4RX — ISIS-FGFR4RX administered subcutaneously
  Other Names: ISIS 463588
  Arms: ISIS-FGFR4RX
Drug: Placebo — Placebo administered subcutaneously
  Arms: Placebo

SUMMARY:
The purpose of this study is to to evaluate the safety, tolerability, pharmacokinetics, and pharmacodynamics of ISIS-FGFR4RX.

ELIGIBILITY:
Inclusion Criteria:

1. Must have given written informed consent (signed and dated) and any authorizations required by local law and be able to comply with all study requirements
2. Male or female patients between the age of 18-65 years, inclusive

   * Females: Must be post-menopausal (defined as 12 months of spontaneous amenorrhea in females > 55 years of age or, in females ≤ 55 years, 12 months of spontaneous amenorrhea without an alternative medical cause and FSH levels in the postmenopausal range for the laboratory involved)
   * Males: Surgically sterile, abstinent or if engaged in sexual relations with women of childbearing potential, patient is utilizing an acceptable contraceptive method during and for 5 months after the last dose of ISIS 463588 or placebo (Study Drug)
3. Body Mass Index (BMI) between 30.0 and 40.0 kg/m2, inclusive
4. Patients who are willing to comply with all scheduled visits, treatment plans, laboratory tests and other study procedures
5. Agree to abstain from alcoholic beverages for at least 48 hours prior to clinic visits
6. Agree to maintain current diet and exercise regimen from Screening until End-of-Study

Exclusion Criteria:

1. Clinically significant abnormalities in medical history (e.g., previous acute coronary syndrome within 6 months of Screening, major surgery within 3 months of Screening) or physical examination
2. Positive test for HIV, hepatitis B or C at Screening
3. Hypothyroidism or Hyperthyroidism
4. Weight change > 5% in the 3 months prior to Screening

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2015-06; Primary Completion 2016-07 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Energy Expenditure using both room calorimetry and hood (metabolic cart) calorimetry | From baseline to the average of weeks 14 and 16
  As measured by:
  * Resting Metabolic rate (kcal/min)
  * Resting metabolic rate adjusted for changes in body composition (kcal/min)
  * Resting fat oxidation (grams/24 hr)

SECONDARY OUTCOMES:
Safety and Tolerability will be assessed by determining the incidence, and severity of adverse effects and changes in laboratory evaluations within each treatment group. | 33 weeks
  Safety results in patients dosed with ISIS 463588 will be compared with those from patients dosed with placebo

CONTACTS AND LOCATIONS:
Locations (1):
- Translational Research Institute for Metabolism and Diabetes, Orlando, Florida, United States